CLINICAL TRIAL: NCT01789515
Title: Diverting Stoma and Postoperative Morbidity After Low Anterior Resection for Rectal Cancer Within an Enhanced Recovery After Surgery,ERAS, Program
Brief Title: Defunctioning Stoma and Postoperative Morbidity
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Kajsa Anderin, Principal Investigator, Karolinska Institutet
Other Study IDs: 2012/538-31/1
Record Dates: First submitted 2012-09-28; First posted 2013-02-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Loopileostomy; Fast Track Program,(Enhanced Recovery After Surgery (ERAS))

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rectal cancer: Low Anterior Resection for Rectal Cancer

SUMMARY:
In an attempt to reduce the risk for anastomotic leakage after low anterior resection it is common to create a diverting stoma at the same procedure. Several studies have shown that ERAS (Enhanced Recovery After Surgery)application reduces the risk of surgical stress and postoperative complications after major colorectal surgery. The aim of this study is to evaluate wether a diverting stoma, after low anterior resection for rectal cancer, affects postoperative morbidity in patients treated within an ERAS program.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* all patients operated with low anterior resection for rectal cancer at Ersta Hospital between 2002 and 2011 registrated in ERAS database

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical anastomotic leakage | 0 to 9 years after surgery
  Evaluate if a diverting stoma after low anterior resection affects postoperative Morbidity in patients treaated within an ERAS program

SECONDARY OUTCOMES:
Permanent stoma | 0 to 9 years after surgery

OTHER OUTCOMES:
Total days of hospital stay | 0-9 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Anderin, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Sweden